CLINICAL TRIAL: NCT04416425
Title: Hemodynamic Change of Coronary Atherosclerotic Plaque After Evolocumab Treatment: A Serial Follow-Up Study by Computed Tomography-Derived Fractional Flow Reserve
Brief Title: Hemodynamic Change of Coronary Atherosclerotic Plaque After Evolocumab Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zibo Central Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZiboCH
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2020-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled Cohort: 200 selected patients will be recruited, who have diagnosed with coronary atherosclerosis disease(stenotic extent from 50% to 69% on major epicardial arteries) by coronary computed tomography angiography(CCTA). Every two weeks, these patients will be treated with Elococumab Injection (1ml:140mg),ih.This therapy will last for one year.

SUMMARY:
Compelling evidences indicate that lipid-lowering therapy can reduce the high-risk plaque feathers and improve the coronary flow reserve. This study is going to investigate the change of lesion-specific hemodynamic significance as determined by ML(Machine Learning)-based CT-FFR (Computed Tomography-Fractional Flow Reserve)after Evolocumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.baseline CCTA revealed at least one lesion with stenotic extent from 50% to 69% on major epicardial arteries (diameter ≧2 mm);
* 2.patients were referred for optimal medical treatment;
* 3.patients agreed to undergo follow-up CCTA at 1-year interval.

Exclusion Criteria:

* 1.patients had previous history of myocardial infarction or coronary revascularization;
* 2.patients were contraindicated to the usage of iodine contrast media;
* 3.image quality of baseline or follow-up CCTA was severely impaired (in presence of severe artifact, non-diagnostic);
* 4.patients withdrew the informed consents during follow-up;
* 5.patients experienced major adverse cardiac events during follow-up;
* 6.patients refused to undergo follow-up CCTA;
* 7.lost follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 200 eligible coronary atherosclerosis disease patients were anticipated to include in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-27 (Estimated)

PRIMARY OUTCOMES:
the change of lesion-specific CT-FFR | June 2020 to December 2021
  After one year's treatment of Elovocumab Injection, the patients will undergo follow-up CCTA again. We will measure the proximal and distal CT-FFR for each lesion.At the same time ,we will calculated the change in CT-FFR value across the lesion(ΔCT-FFR=CT-FFRproximal-CT-FFRdistal).To compare the parameters above,we shall identify whether the treatment of Elovocumab Injection improves the lesion-specific CT-FFR.

OTHER OUTCOMES:
the change of minimal lumen diameter between baseline and follow-up CCTA | June 2020 to December 2021
  After one year's treatment of Elovocumab Injection, the patients will undergo follow-up CCTA again. We will measure the minimal lumen diameter for each lesion. Minimal lumen diameter will be manually measured with a digital caliper at the narrowest level of the lesion using the crosssectional images accroding to the CCTA findings. The results of the minimal lumen diameter at baseline will be compared with results obtained during follow-up to examine the effects of Elovocumab Injection therapy.
the change of total plaque volume (TPV) between baseline and follow-up CCTA | June 2020 to December 2021
  After one year's treatment of Elovocumab Injection, the patients will undergo follow-up CCTA again. We will measure TPV for each lesion. Total plaque volume will be automatically measured using the dedicated plaque analysis software. The results of TPV at baseline will be compared with results obtained during follow-up to examine the effects of Elovocumab Injection therapy.
the change of lesion length between baseline and follow-up CCTA | June 2020 to December 2021
  After one year's treatment of Elovocumab Injection, the patients will undergo follow-up CCTA again. The length of lesion at baseline will be compared with results obtained during follow-up to examine the effects of Elovocumab Injection therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Li, Doctor, Principal Investigator — Zibo Central Hospital
Locations (1):
- Zibo Central Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided